CLINICAL TRIAL: NCT06706336
Title: Radon Asthma Intervention Trial
Acronym: ROME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Wanda Phipatanakul, S Jean Emans, MD Professor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P00050180
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Radon Mitigation (Active Comparator): Active radon mitigation system
  Interventions: Other: radon mitigation system
- Inactive radon mitigation system control( sham) (Sham Comparator): Inactive radon mitigation system looks and sounds like active but doesn't reduce radon ( sham)
  Interventions: Other: Sham (No Treatment)

INTERVENTIONS:
Other: radon mitigation system — standard radon mitigation system used to reduce radon in homes
  Arms: Active Radon Mitigation
Other: Sham (No Treatment) — inactive radon mitigation system
  Arms: Inactive radon mitigation system control( sham)

SUMMARY:
To determine if radon mitigation can improve asthma

DETAILED DESCRIPTION:
We will conduct a randomized, double-blind, sham controlled trial to investigate the efficacy of radon mitigation in the homes of susceptible individuals to provide evidence for health benefits by improving indoor air quality. The trial will include 180 children with asthma. We will install a standard radon specific mitigation system in the participant's home. Health outcomes will be followed over 48 weeks to determine the outcomes of the intervention versus inactive (sham) control.

ELIGIBILITY:
1. Have physician-diagnosed asthma at least 1 year prior to the screening visit
2. Have evidence of uncontrolled disease as defined by at least one of the following:

Use of an asthma medication during the prior 12 months, report of asthma symptoms over the prior 12 months (wheezing/whistling in the chest)(3)

OR

One or more asthma-related hospitalization, emergency room visit

OR

Unscheduled clinic or urgent care facility visit resulting in a burst of systemic steroids (3 days or more of prednisone or equivalent; 1 or more doses of dexamethasone) in the previous 12 months

Exclusion Criteria

1. Not residing at the household for at least 5 days a week or family planning to move from the current home within the next twelve months, or homes with active radon mitigation systems (if home uses a HEPA filter air purifier, family must agree to disable the purifier for 28 days prior to randomization).
2. Lung disease, other than asthma, that requires daily medication (inflammatory diseases, chronic lung diseases aside from asthma, congenital cardiopulmonary conditions requiring medication or surgical treatment),
3. Homes with active HEPA filters will be excluded (even though the role of HEPA filters on radon and radon particles s is expected to be minimum and other exposures can be adjust for in the analysis)
4. Cardiovascular disease that requires daily medication, excluding hypertension
5. Taking a beta-blocker
6. Currently receiving unstable level of Immunotherapy (allergy shots)
7. Coordinator/PI judgment
8. Inability to perform lung function testing
9. Intake of abuse drugs or alcohol, have psychiatric disorders or severe mental disability that interferes with answering questions or following instructions.

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Asthma symptoms | past 2 weeks
  Number of Days With Asthma Symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Wanda Phipatanakul, Principal Investigator — Boston Children's Hospital

IPD SHARING:
Plan to Share IPD: No